CLINICAL TRIAL: NCT00450255
Title: A Phase 2 Study Evaluating the Efficacy of VEGF Trap in Patients With Recurrent Inoperable Stage III or Stage IV Melanoma
Brief Title: VEGF Trap in Treating Patients With Recurrent Stage III or Stage IV Melanoma That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00182; NCI-2009-00182 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHII-77; CDR0000535719; PHII-77 (Other: City of Hope); 7522 (Other: CTEP); N01CM62209 (NIH); P30CA033572 (NIH)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Results first posted 2015-02-04 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-04

CONDITIONS: Ciliary Body and Choroid Melanoma, Medium/Large Size; Extraocular Extension Melanoma; Iris Melanoma; Metastatic Intraocular Melanoma; Recurrent Intraocular Melanoma; Recurrent Melanoma; Stage III Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — aflibercept

ARMS (1):
- Arm I (Experimental): Patients receive Aflibercept IV at 4 mg/kg over 1 hour on day 1. Treatment repeats every 14 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: ziv-aflibercept; Other: pharmacological study

INTERVENTIONS:
Biological: ziv-aflibercept — Given IV
  Other Names: aflibercept; vascular endothelial growth factor trap; VEGF Trap; Zaltrap
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase II trial is studying how well VEGF Trap works in treating patients with recurrent stage III or stage IV melanoma that cannot be removed by surgery. Combinations of biological substances in VEGF Trap may be able to carry tumor-killing substances directly to melanoma cells. It may also stop the growth of melanoma by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the antitumor response rate (complete and partial response) in patients with recurrent inoperable stage III or IV melanoma treated with VEGF Trap.

II. Compare the progression-free survival of patients treated with this regimen vs historical controls.

SECONDARY OBJECTIVES:

I. Determine the overall survival of patients treated with this regimen. II. Determine the toxicity and tolerability of this regimen in these patients. III. Determine the impact of this regimen on laboratory correlates including anti-VEGF Trap antibody testing and pharmacokinetics in these patients.

OUTLINE: This is a multicenter study.

Patients receive VEGF Trap IV over 1 hour on day 1. Treatment repeats every 14 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline, prior to course 2, and 60 days after completion of study treatment for pharmacokinetic and pharmacodynamic studies. Samples are analyzed by enzyme-linked immunosorbent assay.

After completion of study treatment, patients are followed periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage III or IV melanoma
* Cutaneous, ocular, or mucosal melanoma allowed
* Recurrent, inoperable disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* No evidence of CNS disease, including primary brain tumor or brain metastases
* No brain metastases by MRI or CT scan within the past 4 weeks
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 3 months
* WBC ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 75,000/mm³
* Bilirubin < 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* Urine protein:creatinine ratio < 1 OR urine protein < 500 mg by 24-hour urine collection
* PT INR ≤ 1.5 unless on full-dose warfarin
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study treatment
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to agents used in the study
* No serious or nonhealing wound, ulcer, or bone fracture
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* No significant traumatic injury within the past 28 days
* No clinically significant cardiovascular disease, including any of the following:

  * Cerebrovascular accident within the past 6 months
  * Uncontrolled hypertension, defined as blood pressure (BP) > 150/100 mm Hg or systolic BP > 180 mm Hg if diastolic BP < 90 mm Hg within the past 3 months
  * Myocardial infarction, coronary artery bypass graft, or unstable angina within the past 6 months
  * New York Heart Association class III-IV congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Unstable angina pectoris within the past 6 months
  * Clinically significant peripheral vascular disease within the past 6 months
  * Pulmonary embolism, deep vein thrombosis, or other thromboembolic event within the past 6 months
  * No evidence of bleeding diathesis or coagulopathy
* No concurrent uncontrolled illness, including, but not limited to any of the following:

  * Ongoing or active infection
  * Psychiatric illness or social situation that would preclude study compliance
* Recovered from all prior therapy and major surgery
* No prior chemotherapy or hormonal therapy
* More than 7 days since prior core visceral organ biopsy
* More than 4 weeks since prior biologic therapy or radiotherapy
* More than 28 days since prior major surgery or open biopsy
* No concurrent major surgery
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* Concurrent full-dose warfarin with PT INR > 1.5 allowed provided the following criteria are met:

  * INR in range (2-3) on a stable dose of oral anticoagulant or low molecular weight heparin
  * No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Tarhini, Principal Investigator — University of Pittsburgh
Locations (1):
- City of Hope, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I
Started | 41
Completed | 40
Not Completed | 1
Not completed — Prior RFA ablation of liver | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 41
Age, Continuous [Median (Full Range); unit: years] | 57 [23 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 26
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 41
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (CR + PR)
Description: Using the RECIST v1.0 criteria for target lesions assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response = CR + PR.",
Time Frame: Start of treatment to disease progression/recurrence, up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm I: Patients receive Aflibercept IV at 4 mg/kg 1 hour on day 1. Treatment repeats every 14 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.
  ziv-aflibercept: Given IV
  pharmacological study: Correlative studies
Arm/Group | Arm I
Number analyzed (Participants) | 40
percentage of participants | 7.5 [2 to 20]

2. Primary Outcome: 4 Month Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 4 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm I
Number analyzed (Participants) | 40
percentage of patients | 50 [34 to 66]

3. Secondary Outcome: Overall Survival
Description: Will be estimated by the Kaplan-Meier method.
Time Frame: From the initial date of treatment to the recorded date of death, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I
Number analyzed (Participants) | 40
Months | 16.3 [9.2 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

4. Secondary Outcome: Number of Participants With Toxicities
Description: The descriptions and grading scales found in the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 were utilized for AE grading and reporting. Grade 3 and higher adverse events considered possibly, probably or definitely related to aflibercept are summarized.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 41
Participants
  Grade 3 : Thrombocytopenia | 1
  Grade 3 : Hypertension | 9
  Grade 3 : Hypotension | 1
  Grade 3 : LV Diastolic Dys | 1
  Grade 3 : GI Bleed | 1
  Grade 3 : Cerebrovascular ischemia | 0
  Grade 3 : Headache | 1
  Grade 3 : Extraocular muscle paresis | 1
  Grade 3 : Fatigue | 1
  Grade 3 : Hyponatremia | 2
  Grade 3 : Osteonecrosis of mandibular bone | 1
  Grade 3 : Back Pain | 1
  Grade 3 : Chest Pain | 1
  Grade 3 : Increased creatinine | 1
  Grade 3 : Proteinuria | 6
  Grade 4 : Thrombocytopenia | 0
  Grade 4 : Hypertension | 0
  Grade 4 : Hypotension | 0
  Grade 4 : LV Diastolic Dys | 0
  Grade 4 : GI Bleed | 0
  Grade 4 : Cerebrovascular ischemia | 1
  Grade 4 : Headache | 0
  Grade 4 : Extraocular muscle paresis | 0
  Grade 4 : Fatigue | 0
  Grade 4 : Hyponatremia | 0
  Grade 4 : Osteonecrosis of mandibular bone | 0
  Grade 4 : Back Pain | 0
  Grade 4 : Chest Pain | 0
  Grade 4 : Increased creatinine | 0
  Grade 4 : Proteinuria | 0

5. Secondary Outcome: Impact of the VEGF Trap Therapy on Laboratory Correlates
Time Frame: Up to 5 years
Population: Laboratory Correlate data were not collected.
Arm/Group | Arm I
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events took place over a period of 1 year and 4 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 13/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=41)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Extraocular muscle paresis (Eye disorders) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Peritoneal pain (Gastrointestinal disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Gingival infection (Infections and infestations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=41)
Hemoglobin decreased (Blood and lymphatic system disorders) | 6 (9)
Atrial fibrillation (Cardiac disorders) | 1 (4)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (3)
External ear pain (Ear and labyrinth disorders) | 1 (1)
Hearing loss (Ear and labyrinth disorders) | 1 (2)
Hearing test abnormal (Ear and labyrinth disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (2)
Photophobia (Eye disorders) | 1 (2)
Vision blurred (Eye disorders) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 8 (13)
Constipation (Gastrointestinal disorders) | 7 (9)
Diarrhea (Gastrointestinal disorders) | 6 (7)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 3 (6)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (3)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 12 (18)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 9 (13)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (2)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (10)
Chest pain (General disorders) | 2 (4)
Chills (General disorders) | 1 (1)
Disease progression (General disorders) | 23 (23)
Edema limbs (General disorders) | 10 (18)
Facial pain (General disorders) | 2 (3)
Fatigue (General disorders) | 23 (37)
Fever (General disorders) | 3 (4)
General symptom (General disorders) | 1 (2)
Localized edema (General disorders) | 1 (1)
Pain (General disorders) | 7 (26)
Immune system disorder (Immune system disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Gingival infection (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 4 (5)
Sinusitis (Infections and infestations) | 5 (7)
Skin infection (Infections and infestations) | 2 (2)
Tooth infection (Infections and infestations) | 3 (4)
Upper aerodigestive tract infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (4)
Vaginal infection (Infections and infestations) | 1 (1)
Intraoperative respiratory injury - Nasal cavity (Injury, poisoning and procedural complications) | 1 (1)
Stomal ulcer (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 10 (23)
Alkaline phosphatase increased (Investigations) | 12 (26)
Aspartate aminotransferase increased (Investigations) | 13 (37)
Bilirubin increased (Investigations) | 2 (9)
Creatine phosphokinase increased (Investigations) | 2 (5)
Creatinine increased (Investigations) | 9 (18)
Laboratory test abnormal (Investigations) | 9 (21)
Leukocyte count decreased (Investigations) | 1 (2)
Lymphocyte count decreased (Investigations) | 8 (21)
Neutrophil count decreased (Investigations) | 1 (4)
Platelet count decreased (Investigations) | 3 (7)
Weight loss (Investigations) | 4 (6)
Anorexia (Metabolism and nutrition disorders) | 5 (6)
Blood glucose increased (Metabolism and nutrition disorders) | 10 (34)
Serum albumin decreased (Metabolism and nutrition disorders) | 5 (13)
Serum calcium decreased (Metabolism and nutrition disorders) | 3 (4)
Serum glucose decreased (Metabolism and nutrition disorders) | 2 (3)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 8 (12)
Serum sodium decreased (Metabolism and nutrition disorders) | 14 (32)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Joint pain (Musculoskeletal and connective tissue disorders) | 8 (12)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (11)
Upper extremity dysfunction (Musculoskeletal and connective tissue disorders) | 1 (3)
Dizziness (Nervous system disorders) | 6 (8)
Headache (Nervous system disorders) | 21 (37)
Nystagmus (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Sinus pain (Nervous system disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 3 (3)
Agitation (Psychiatric disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 2 (3)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 7 (11)
Glomerular filtration rate decreased (Renal and urinary disorders) | 1 (1)
Hemoglobin urine positive (Renal and urinary disorders) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 2 (6)
Protein urine positive (Renal and urinary disorders) | 13 (34)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1)
Uterine hemorrhage (Reproductive system and breast disorders) | 1 (3)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (17)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 10 (21)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (25)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 13 (30)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash desquamating (Skin and subcutaneous tissue disorders) | 9 (12)
Skin disorder (Skin and subcutaneous tissue disorders) | 5 (22)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (4)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2)
Sweating (Skin and subcutaneous tissue disorders) | 5 (6)
Flushing (Vascular disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 30 (55)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less